CLINICAL TRIAL: NCT06515951
Title: Diagnostic Accuracy of the STANDING Algorithm for the Differential Diagnosis of Vertigo in the Emergency Department: a Multicenter Study.
Brief Title: Effectiveness of the STANDING Algorithm for the Differential Diagnosis of Vertigo
Acronym: STANDING-M
Status: Completed | Type: Observational
Sponsor: Peiman Nazerian (Other)
Collaborators: Ospedale San Giuseppe di Empoli (Other); Ospedale Santo Stefano (Other); Azienda USL Toscana Nord Ovest (Other); Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Sponsor-Investigator, Peiman Nazerian, Medical Doctor, Azienda Ospedaliero-Universitaria Careggi
Organization: Azienda Ospedaliero-Universitaria Careggi (Other)
Other Study IDs: 11085
Record Dates: First submitted 2023-05-10; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Vertigo
Keywords: Central vertigo; Peripheral vertigo; Ischemic stroke
MeSH Terms: conditions — Vertigo; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STANDING group: Consecutive adult patients who access the emergency room due to vertigo / imbalance will be considered eligible for the study. in this group patients will be evaluated by STANDING protocol
  Interventions: Diagnostic Test: STANDING algorithm
- Control group: Consecutive adult patients who access the emergency room due to vertigo / imbalance will be considered eligible for the study. in this group patients will be evaluated by standard of care

INTERVENTIONS:
Diagnostic Test: STANDING algorithm — The STANDING algorithm is composed by four steps. The first phase consists in evaluating the presence of spontaneous nystagmus at rest for at least five minutes with and without Frenzel goggles in order to assess if a acute vestibular syndrome is present. If there is not a spontaneous nystagmus, then positional maneuvers (Pagnini-Mc Cure and Dix-Hallpike) have to be performed. Otherwise if spontaneous nystagmus is observed, its feature are fundamental to diagnose a central vertigo. If nystagmus characteristics suggest a peripheral form, the head impulse test is performed by instructing the patient to keep eyes on a fixed target and then turned the head quickly. An abnormal response is typical of vestibular neuritis. In any cases after the described maneuvers, the patient must be evaluated when standing up and walking: if this turn out to be impossibile, the test is indicative of central nervous system disease.
  Groups: STANDING group

SUMMARY:
Differential diagnosis of vertigo is complex especially in emergency department, nevertheless it is crucial. The aim of this study is to assess the accuracy of STANDING algorithm for discriminate central from peripheral type of vertigo, identifying more easily the presence of ischemic stroke.

DETAILED DESCRIPTION:
Vertigo represents a common medical problem which afflicts about 20-30% of the population and it is a frequent cause of abstention from work and disability. In most cases it is provoked by a benign disease of inner ear, however it can be the main symptom of a more dangerous illness like ischemic or hemorragic stroke, cerebral neoplasm or demyelinating disease. Indeed, vertigo is the prevailing clinical problem in patients with misdiagnosed ischemic stroke, leading to an increase of mortality in the acute phase of disease. In the current state, two diagnostic algorithm have been proposed for the evaluation of acute vertigo, named with the acronyms HINTS and STANDING. The former is characterized by high sensibility and specificity when utilized by a specialist physician, but it is cumbersome to used in emergency department. Conversely, the latter has been validated exactly in this setting and comprises the evaluation of benign paroxysmal positional vertigo and of upright position. The aim of this study is to estimate the accuracy of STANDING algorithm in differentiating peripheral vertigo from central from, in particular ischemic stroke, and its potential usefulness in decreasing the use of neuroimaging and specialist consultant.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age.
* patients affected by vertigo, dizziness or balance disorder.

Exclusion Criteria:

* age under 18.
* patients unable to cooperate (with severe dementia or incapable to provide consensus).
* patients affected by disease of cervical spine or any trauma of this part of body that contraindicate the manipulation of neck.
* impractical follow-up.
* dying patient (less three estimated months to live).
* patients with neurologic deficit identified during triage examination (Cincinnati Prehospital stroke scale, CPSS>0) of suffering from another disease that can be the cause of dizziness/balance disorder (e.g. anemia, arrhythmia, hypoglycemia, alcoholic intoxication).
* patients without symptoms at the time of examination.
* patients who deny the participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every adult patient presenting in emergency department with vertigo, dizziness or balance disorder.
Sampling Method: Probability Sample
Enrollment: 456 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of STANDING algorithm for the diagnosis of types of vertigo. | Thirty days
  Accuracy (proportion of true positive and negative cases among the total number of cases examined) together with sensitivity, specificity, negative and positive predictive values, negative and positive likelihood ratios of STANDING algorithm performed by emergency physicians to distinguish central and peripheral vertigo.

SECONDARY OUTCOMES:
Change in the use of neuroimaging | Thirty days
  Evaluation if the use of STANDING algorithm can reduce the number neuroimaging (a composite of CT of the head and brain MRI) exams performed in patients with suspected central vertigo according to the STANDING algorithm.
Safety of hospital discharge | Thirty days
  Evaluation if the use of STANDING algorithm allows a safe discharge of patients with diagnosis of benign vertigo. At 1 month follow-up we evaluate the composite of: number of readmissions for stroke, need for cerebral revasculation procedures, for neurosurgery or all cause death or death for stroke) in patients without suspected central vertigo according to the STANDING algorithm.
Accuracy for diagnosis of stroke | Thirty days
  Accuracy (proportion of true positive and negative cases of stroke among the total number of cases examined)
Change in the use of specialist consultant | thirty days
  Evaluation if the use of STANDING algorithm can reduce the number of specialist medical consultations (composite of neurological and ENT consultations) performed in patients with suspected central vertigo according to the STANDING algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Magazzini, MD, Study Chair — Direttore Dipartimento Emergenza Urgenza e Area Critica AUTC; Maurizio Bartolucci, MD, Study Chair — Direttore Dipartimento Diagnostica per immagini AUTC; Paola Bartalucci, MD, Study Chair — Medicina d'Urgenza Empoli AUTC; Claudia Casula, MD, Study Chair — Medicina d'Urgenza Empoli AUTC; Simone Vanni, MD, Principal Investigator — Direttore SOC Medicina d'Urgenza EMPOLI; Direttore Area della Formazione Dipartimento Emergenza Urgenza e Area Critica AUTC
Locations (4):
- Italy (4):
  - Azienda USL Toscana Centro, Medicina d'Urgenza e Dipartimento Emergenza e Area Critica, Empoli, Firenze
  - Ospedale Versilia, Medicina d'Urgenza, Viareggio, Lucca
  - Azienda Ospedaliera Universitaria Careggi, Medicina d'Urgenza, Florence, Tuscany
  - Nuovo Ospedale di Prato, Medicina d'Urgenza, Prato

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Validation STANDING study, monocentric — https://www.frontiersin.org/articles/10.3389/fneur.2017.00590/full
- See also: Derivation STANDING study, monocentric — https://www.actaitalica.it/issues/2014/6-2014/08-Vanni.pdf